CLINICAL TRIAL: NCT00096239
Title: Phase II Open-Label, Multi-Center Study of CP-547, 632, an Oral Tyrosine Kinase Inhibitor of VEGFR-2, in Subjects With Recurrent or Persistent Small-Volume Epithelial Ovarian Cancer, Primary Peritoneal Serous Cancer, or Fallopian Tube Cancer
Brief Title: CP-547,632 in Treating Patients With Recurrent or Persistent Ovarian Cancer, Primary Peritoneal Cancer, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000390237; UCLA-0311057-01; PFIZER-A3521003
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2005-02

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; primary peritoneal cavity cancer; fallopian tube cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — 3-(4-bromo-2,6-difluorobenzyloxy)-5-(3-(4-pyrrolidin-1-ylbutyl)ureido)isothiazole-4-carboxylic acid amide

INTERVENTIONS:
Drug: CP-547,632

SUMMARY:
RATIONALE: CP-547,632 may stop the growth of tumor cells by blocking the enzymes necessary for their growth and by stopping blood flow to the tumor.

PURPOSE: This phase II trial is studying how well CP-547,632 works in treating patients with recurrent or persistent ovarian cancer, primary peritoneal cancer, or fallopian tube cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of CP-547,632, in terms of clinical response benefit (CA 125 response [complete response (CR) or partial response (PR)] or stable disease ≥ 16 weeks), in patients with recurrent or persistent small-volume ovarian epithelial, primary peritoneal serous, or fallopian tube cancer.

Secondary

* Determine progression-free survival of patients treated with this drug.
* Determine CA 125 response (CR or PR) rate in patients treated with this drug.
* Determine duration of CA 125 response in patients treated with this drug.
* Determine the safety of this drug in these patients.
* Correlate the steady state plasma concentration of this drug with efficacy and toxicity in these patients.
* Correlate clinical outcome with an angiogenic profile derived from measurement of serum vascular endothelial growth factor, basic fibroblast growth factor, and interleukin-8 in patients treated with this drug.
* Determine changes in the Hospital Anxiety and Depression Scale (HADS) in patients treated with this drug.

OUTLINE: This is an open-label, multicenter study.

Patients receive oral CP-547,632 once daily on days 1-28. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 30 days and then every 3 months for 2 years.

PROJECTED ACCRUAL: A total of 10-29 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial, primary peritoneal serous, or fallopian tube cancer

  * Recurrent or persistent disease

    * Elevated CA 125, defined as ≥ 40 U/mL on 2 separate consecutive measurements taken ≥ 1 week apart
* No definitive disease OR small-volume disease (≤ 2 cm by spiral or conventional CT scan or clinical exam)
* Asymptomatic disease

PATIENT CHARACTERISTICS:

Age

* 26 and over (age 18 to 25 allowed provided there is closure of the epiphyses on radiography)

Performance status

* ECOG 0-1

Life expectancy

* More than 6 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* No bleeding disorders
* No hemorrhage ≥ grade 2 within the past 12 months

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* ALT and/or AST ≤ 2.5 times ULN
* Albumin ≥ 3.2 g/dL
* PT/PTT ≤ 1.5 times ULN
* INR ≤ 1.5

Renal

* Creatinine ≤ 1.5 times ULN OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* QTc ≤ 460 msec by ECG
* No unstable angina within the past 6 months
* No decompensated congestive heart failure within the past 6 months
* No myocardial infarction within the past 6 months
* No serious cardiac arrhythmias or conduction abnormalities, including any history of recurrent ventricular arrhythmia, within the past 6 months
* No cardiomyopathy
* No history of syncope associated with arrhythmia
* No uncontrolled hypertension within the past 3 weeks, defined as systolic blood pressure > 150 mm Hg or diastolic blood pressure > 90 mm Hg on ≥ 2 of 3 blood pressure readings taken ≥ 5 minutes apart
* No thrombotic cardiovascular events, including transient ischemic attacks, within the past 12 months

Gastrointestinal

* Able to take oral medication
* No malabsorption syndromes
* No active gastrointestinal bleeding (hematemesis, hematochezia, or melena), unrelated to cancer, within the past 3 months
* No requirement for IV alimentation

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No active infection
* No uncontrolled diabetes
* No dementia, altered mental status, or uncontrolled psychiatric illness that would preclude giving informed consent or study compliance
* No other serious uncontrolled medical disorder that would preclude study participation
* No other active malignancy within the past 3 years except treated limited stage basal cell or squamous cell skin cancer or carcinoma in situ of the breast or cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior exposure to mouse antibodies
* No prior vascular endothelial growth factor (VEGF) or VEGF-receptor targeted therapy
* No other prior antiangiogenic anticancer therapy, including thalidomide
* No concurrent prophylactic colony-stimulating factors (i.e., filgrastim [G-CSF] or sargramostim [GM-CSF])
* No concurrent immunotherapy

Chemotherapy

* Prior chemotherapy allowed provided patient received only a first-line platinum-based chemotherapy regimen with or without systemic consolidation chemotherapy
* At least 3 weeks since prior chemotherapy and recovered (excluding alopecia)
* No concurrent chemotherapy

Endocrine therapy

* At least 3 weeks since prior hormonal therapy for ovarian cancer and recovered
* Concurrent hormone replacement therapy allowed
* No concurrent chronic oral or IV corticosteroids
* No concurrent hormonal therapy, including tamoxifen

Radiotherapy

* No concurrent radiotherapy

Surgery

* More than 4 weeks since prior major surgical procedure
* No prior gastric resection

Other

* More than 3 weeks since prior investigational therapy
* More than 4 weeks since prior major medical interference with the peritoneum or pleura
* More than 3 months since prior treatment for active ulcer disease
* No prior consolidation intraperitoneal therapy using cytotoxic agents for ovarian cancer
* No concurrent antiarrhythmics

  * Beta blockers or calcium channel blockers used for other indications allowed
* No concurrent grapefruit juice
* No concurrent therapeutic anticoagulant therapy or chronic daily aspirin > 325 mg/day

  * Concurrent low-dose anticoagulants for maintenance of central venous access allowed
* No other concurrent experimental or anticancer therapy for the primary disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-12; Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. Pegram, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States